CLINICAL TRIAL: NCT06108986
Title: Effects of Tabata Training Versus Plyometric Training on Range of Motion of ap Chagi, Agility and Vertical Jump in Taekwondo Players
Brief Title: Tabata vs Plyometric Training on Range of Motion, Agility and Vertical Jump in Taekwondo Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0441
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: High-Intensity Interval Training; Plyometric Exercise; Martial Arts
Keywords: Tabata training; Plyometric training; Taekwondo
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: randomized clinical trail
Who Masked: Outcomes Assessor
Masking Description: the assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tabata training (Experimental): Group A will perform tabata that includes squats, push up, side jump, medicine ball pass, commando dance, plank, skip rope, burpees. three sessions per week for six weeks.
  Interventions: Other: tabata training
- plyometric training (Experimental): Group B will perform plyometric training that includes squats, ankle hopes, jumps in a place, lunges, shuffling, stair jump exercises. three sets of eight reps, three sessions per week for six weeks.
  Interventions: Other: plyometric training

INTERVENTIONS:
Other: tabata training — this include tabata training thrice a week for six weeks
  Arms: tabata training
Other: plyometric training — this include plyometric training thrice a week for six weeks
  Arms: plyometric training

SUMMARY:
The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah Internatinal University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Subjects in Group A will receive tabata training. Group B will receive plyometric training.

DETAILED DESCRIPTION:
the objective of the study is to determine the effects of tabata training versus plyometric training on range of motion of ap chagi, agility and vertical jump in taekwondo players. The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah Internatinal University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Subjects in Group A will receive tabata training. Group B will receive plyometric training. The outcome measures will be assessed by goniometrer, quadrant jump test - agility and vertical jump test.

The data will be analyzed by SPSS, version 25. Statistical significance is P= 0.05.

ELIGIBILITY:
Inclusion Criteria:

Taekwondo players, Both male and female players., Players aged 12- 25 years, Players who are playing taekwondo from at least past six months, Individuals with BMI between 18.5- 24.9

Exclusion Criteria:

Out of practice players, Players with any musculoskeletal injury within past four weeks, Unwilling participants, Players with any systemic disease

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
range of motion | pre and 6 weeks post interventional
  range of motion of ap chagi will be measured by goniometer
agility | pre and 6 weeks post interventional
  Quadrant jump test - agility is used to measure agility
vertical jump | pre and 6 weeks post interventional
  vertical jump test is use to measure lower extremity power

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Basim, DPT, Principal Investigator — Study Principal Investigator
Locations (1):
- Yaldarm taekwondo Academy, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li B, Ding C, Fan F, Shi H, Guo L, Yang F. Associations Between Psychological Profiles and Performance Success Among Professional Taekwondo Athletes in China: A Multidimensional Scaling Profile Analysis. Front Psychol. 2020 May 15;11:822. doi: 10.3389/fpsyg.2020.00822. eCollection 2020. PMID 32499737
- [Background] Norjali Wazir MRW, Van Hiel M, Mostaert M, Deconinck FJA, Pion J, Lenoir M. Identification of elite performance characteristics in a small sample of taekwondo athletes. PLoS One. 2019 May 31;14(5):e0217358. doi: 10.1371/journal.pone.0217358. eCollection 2019. PMID 31150424
- [Background] Jlid MC, Racil G, Coquart J, Paillard T, Bisciotti GN, Chamari K. Multidirectional Plyometric Training: Very Efficient Way to Improve Vertical Jump Performance, Change of Direction Performance and Dynamic Postural Control in Young Soccer Players. Front Physiol. 2019 Dec 9;10:1462. doi: 10.3389/fphys.2019.01462. eCollection 2019. PMID 31920686
- [Background] Cherni Y, Jlid MC, Mehrez H, Shephard RJ, Paillard T, Chelly MS, Hermassi S. Eight Weeks of Plyometric Training Improves Ability to Change Direction and Dynamic Postural Control in Female Basketball Players. Front Physiol. 2019 Jun 13;10:726. doi: 10.3389/fphys.2019.00726. eCollection 2019. PMID 31263427
- [Background] Viana RB, de Lira CAB, Naves JPA, Coswig VS, Del Vecchio FB, Gentil P. Tabata protocol: a review of its application, variations and outcomes. Clin Physiol Funct Imaging. 2019 Jan;39(1):1-8. doi: 10.1111/cpf.12513. Epub 2018 Apr 2. PMID 29608238
- [Background] Tabata I. Tabata training: one of the most energetically effective high-intensity intermittent training methods. J Physiol Sci. 2019 Jul;69(4):559-572. doi: 10.1007/s12576-019-00676-7. Epub 2019 Apr 19. PMID 31004287